CLINICAL TRIAL: NCT02248376
Title: Non-stick Gel Applicated After Scraping Surgery for Natural Miscarriage and Uterine Synechiae Prevention
Brief Title: Hyaluronic Acid and Uterine Synechiae
Acronym: HYFACO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P 130911; AOR13019 (Other: Assistance Publique)
Record Dates: First submitted 2014-09-22; First posted 2014-09-25 (Estimated); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Uterine Synechiae After Scraping for Natural Miscarriage
Keywords: Uterine synechiae Scraping surgery Natural miscarriage
MeSH Terms: interventions — Gels

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gel + (Experimental): Patients aged of more than 18 years-old coming for a natural miscarriage who will have the stick gel application at the end of the scraping surgery.
  Interventions: Drug: Gel
- Gel - (No Intervention): Patients aged of more than 18 years-old coming for a natural miscarriage who will not have the non-stick gel application at the end of the scraping surgery.

INTERVENTIONS:
Drug: Gel — Patients aged of more than 18 years-old coming for a natural miscarriage who will have the stick gel application at the end of the scraping surgery.
  Arms: Gel +

SUMMARY:
The primary purpose of the study is to compare efficiency of a non-stick gel application after scraping surgery for natural miscarriage with no non-stick gel application after scraping surgery.

Post-scraping uterine synechiae rate will be established at the diagnostical hysteroscopy 6-8 weeks after surgery.

DETAILED DESCRIPTION:
Women patients coming for natural miscarriage will be compared according to whether a non-stick gel will be applicated or not after scraping surgery.

6-8 weeks after this surgery uterine synechiae rate will be established at a diagnostical hysteroscopy. Proofreading of this exam will be made by 2 experts at the end of the study without knowing the randomization arm.

Long-term follow-up of the patients will be performed to evaluate the effect of the non-stick gel application on post-surgical fertility at 6, 12, and 24 months after scraping surgery using questionnaire asked by post, mail or phone.

ELIGIBILITY:
Inclusion Criteria:

* Women patients aged between 18 and 46 years old
* Term ≥ 7 weeks amenorrhea and ≤ 14 weeks amenorrhea
* Blighted ovum or not completed miscarriage or haemorrhagic miscarriage or retention miscarriage
* Consent signature
* Social security coverage
* Women who wants to be pregnant

Exclusion Criteria:

* Infected miscarriage
* Uncertain diagnosis between miscarriage and extra-uterine pregnancy
* Hydatiform mole
* Uterine synechiae history
* Surgical zone infection
* Hyalobarrier® gel Endo hypersensitivity
* Clotting disorder
* Unstable diabetes
* Maternal malignant diseases
* Psychiatric disorder
* Incapacity in understanding the consent form and the questionnaires
* Law protected adult person

Ages: 18 Years to 46 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 364 (Actual)
Dates: Start 2014-11-14 (Actual); Primary Completion 2018-09-14 (Actual); Study Completion 2018-09-14 (Actual)

PRIMARY OUTCOMES:
Evaluation of post-surgical uterine synechiae rate during a diagnostical hysteroscopy. | 6-8 weeks after scraping surgery
  Diagnostical hysteroscopy performed 6-8 weeks after scraping surgery.

SECONDARY OUTCOMES:
Evaluation of the effect of the non-stick gel application on the post-surgical fertility 6, 12, and 24 months after scraping surgery. | 6, 12 and 24 months after scraping surgery
  Evaluation using questionnaires asked by post, mail or phone at 6, 12, and 24 months after scraping surgery.
Evaluation of the obstetric complication rate 12 and 24 months after scraping surgery. | Evaluation of the obstetric complication rate 12 and 24 months after scraping surgery.
  Evaluation using questionnaires asked by post, mail or phone at 12 and 24 months after scraping surgery.
Evaluation of post-surgical synechiae stretch and severity | 6-8 weeks after scraping surgery
  Synechiae stretch and severity will be evaluated by the American Fertility Society classification (rAFS).
Consistency assessment between synechiae evaluation performed at the diagnostical hysteroscopy and the synechiae evaluation performed by the 2 experts at the end of the study | 36 months
  Synechiae stretch and severity will be evaluated by the American Fertility Society classification (rAFS).

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis Benifla, MD-PhD, Principal Investigator — Assistance Publique
Locations (1):
- Hôpital Lariboisière - Service de Gynécologie-Obstétrique, Paris, France

REFERENCES:
- [Derived] Sroussi J, Bourret A, Pourcelot AG, Thubert T, Lesavre M, Legendre G, Tuffet S, Rousseau A, Benifla JL; HYFACO group. Does hyaluronic acid gel reduce intrauterine adhesions after dilation and curettage in women with miscarriage? A Multicentric randomized controlled trial (HYFACO Study). Am J Obstet Gynecol. 2022 Oct;227(4):597.e1-597.e8. doi: 10.1016/j.ajog.2022.05.064. Epub 2022 Jun 3. PMID 35667420